CLINICAL TRIAL: NCT05935332
Title: A Phase 2 Study to Evaluate the Efficacy and Safety of RPT193 in Adults With Moderate-to-severe T2-high Asthma Who Are Partially Controlled on Inhaled Corticosteroid and Long-acting Beta 2 Agonist Therapy
Brief Title: Phase 2 Study to Evaluate RPT193 in Adults With Moderate to Severe T2-high Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study on clinical hold by FDA
Sponsor: RAPT Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPT193-03
Record Dates: First submitted 2023-06-26; First posted 2023-07-07 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Asthma
Keywords: asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RPT193 400 mg (Experimental)
  Interventions: Drug: RPT193
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: RPT193 — RPT193 is an antagonist of the C-C motif chemokine receptor 4 (CCR4) that inhibits CCR4-mediated chemotaxis toward both CCL22 and CCL17
  Arms: RPT193 400 mg
Other: Placebo — placebo
  Arms: Placebo

SUMMARY:
Randomized, multi-center, double-blind, placebo-controlled, parallel group, proof of-concept study with RPT193 in subjects with T2-high, moderate-to-severe asthma who are partially controlled on medium or high doses of inhaled corticosteroids (ICS) in combination with long-acting beta 2 agonist (LABA).

DETAILED DESCRIPTION:
Randomized, multi-center, double-blind, placebo-controlled, parallel group, proof of-concept study with RPT193 in subjects with T2-high, moderate-to-severe asthma who are partially controlled on medium or high doses of inhaled corticosteroids (ICS) in combination with long-acting beta 2 agonist (LABA).

After a screening period subjects will receive standardized, inhaled therapy during a run-in period. Subjects will be randomized to receive RPT193 or placebo through Week 14. All enrolled subjects will receive background inhaled therapy with ICS and LABA.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of asthma for ≥6 months
* Pre-bronchodilator FEV1 of >40% and <80%
* History of treatment with corticosteroid or hospitalization for worsening asthma
* Medium- or high-dose inhaled corticosteroid use

Exclusion Criteria:

* History of smoking/vaping
* History of severe COVID
* Serious and/or uncontrolled pulmonary, cardiac, immune system conditions
* Requires systemic oral or IV corticosteroids in the month prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with a Loss of Asthma Control event as defined by criteria listed | 14 weeks
  ≥ 30% reduction in peak expiratory flow; ≥ 6 additional inhalations of short-acting beta 2 agonist; increase by factor of 4 or more of inhaled corticosteroids; and/or evidence of a severe asthma exacerbation

SECONDARY OUTCOMES:
Frequency of treatment-emergent adverse events as assessed by CTCAE v5.0 | 20 weeks
  Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Cheng, MD, PhD, Study Director — RAPT Therapeutics, Inc.
Locations (29):
- United States (13):
  - Allergy and Asthma Associates of Santa Clara Valley Research Center, San Jose, California
  - Bensch Clinical Research LLC, Stockton, California
  - Allianz Research Institute, Westminster, California
  - Allianz Research Institute CO, Aurora, Colorado
  - Sonce Medical Research, Miami, Florida
  - Coral Research Clinical Corp, Miami, Florida
  - San Marcos Research Clinic, Miami Lakes, Florida
  - Clinical Research Trials of Florida, Tampa, Florida
  - OK Clinical Research LLC, Edmond, Oklahoma
  - Velocity Clinical Research Grants Pass, Grants Pass, Oregon
  - Western Sky Medical Research, El Paso, Texas
  - Metroplex Pulmonary & Sleep Center, McKinney, Texas
  - Allergy, Asthma & Sinus Ceneter SC, Greenfield, Wisconsin
- Bulgaria (6):
  - Medical Center "Zadrave-1", Kozloduy
  - Medical Center Excelsior, Sofia
  - Diagnostic-Consultative Center Convex Ltd., Sofia
  - University Multiprofile Hospital for Active Treatment, Stara Zagora
  - Medical Center "ResearchExpert" Ltd, Varna
  - Specialized Hospital for Active Treatment of Pneumo-Phthisiatric Diseases - Vratsa, Vratsa
- MediTrial s.r.o, Jindřichův Hradec, Czechia
- Poland (9):
  - Trialmed Sp z. o.o.o CRS Warszawa, Warsaw, Solipska
  - Centrum Medycyny Oddechowej Mróz Spółka Jawna, Bialystok
  - NZOZ Poradnie Specjalistyczne Atopia, Krakow
  - IP Clinic Sp. z.o.o, Lodz
  - Centrum Diagnostyczno Terapeutyczne MEDICUS Sp. z o.o. - Szpital, Lubin
  - Trialmed CRS (Piotrków Trybunalski), Piotrkow Trybunalski
  - Specjalistyczna Przychodnia Lekarska Alergo-Med sp. z o.o, Poznan
  - Michal Bogacki - Dobrostan, Wroclaw
  - Lekarze Specjaliści - J. Małolepszy i Partnerzy, Wroclaw

IPD SHARING:
Plan to Share IPD: No